CLINICAL TRIAL: NCT03233724
Title: Phase I/II Evaluation of Oral Decitabine/Tetrahydrouridine as Epigenetic Priming for Pembrolizumab Immune Checkpoint Blockade in Inoperable Locally Advanced or Metastatic Non-Small Cell Lung Cancers, Esophageal Carcinomas, or Pleural Mesotheliomas
Brief Title: Oral Decitabine and Tetrahydrouridine as Epigenetic Priming for Pembrolizumab-Mediated Immune Checkpoint Blockade in Patients With Inoperable, or Unresectable Locally Advanced or Metastatic Non-Small Cell Lung Cancers and Esophageal Carcinomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to drug supply issues.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Schrump, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170140; 17-C-0140
Record Dates: First submitted 2017-07-28; First posted 2017-07-31 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Cancer; Non-Small Cell Lung Cancer; Carcinoma, Esophageal; Malignant Pleural Mesotheliomas
Keywords: PD-L1; Demethylating Agents and Histone Deacetylase (HDAC) Inhibitors; DNA Hypomethylating Agent; Cytidine Deaminase; Checkpoint Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Esophageal Neoplasms; Mesothelioma, Malignant | interventions — Decitabine; Tetrahydrouridine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Dose Escalation (Experimental): Decitabine (DAC)-Tetrahydrouridine (THU) + pembrolizumab at escalating doses
  Interventions: Drug: Decitabine (DAC); Drug: Tetrahydrouridine (THU); Drug: Pembrolizumab
- 2/Dose Expansion (Experimental): Decitabine (DAC)-Tetrahydrouridine (THU) + pembrolizumab at the dose established in Arm 1
  Interventions: Drug: Decitabine (DAC); Drug: Tetrahydrouridine (THU); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Decitabine (DAC) — Administered orally on two consecutive days (preferably Tuesday and Wednesday) for two weeks out of three weeks x 9 weeks
  Other Names: Dacogen
Drug: Tetrahydrouridine (THU) — Administered orally on two consecutive days (preferably Tuesday and Wednesday) for two weeks out of three weeks x 9 weeks
Drug: Pembrolizumab — 200 mg intravenous (IV) once a day every Wednesday, Thursday or Friday every 3 weeks.
  Other Names: Keytruda

SUMMARY:
Background:

Non-small cell lung cancer (NSCLC) is the most common type of lung cancer. Lung cancer is the leading cause of cancer-related death in the United States. Most people with lung cancer are already in the advanced stages of the disease by the time they see a doctor. Researchers want to see if combining an approved drug with two new drugs can help.

Objective:

To study if tetrahydrouridine-decitabine (THU-DAC) with pembrolizumab is safe and effective in people with non-small cell lung cancer that cannot be removed by surgery.

Eligibility:

People 18 years and older who have NSCLC that cannot be removed by surgery

Design:

Participants will be screened with

* Medical history
* Physical exam
* Blood and urine tests
* Tests of heart and lung function

They may have a small tumor sample taken (biopsy). They may have tumor scans.

Before starting treatment, participants will repeat the screening tests. They will also give a stool sample.

The study will be done in 3-week cycles for up to 6 cycles.

* Participants will take the 2 study drugs by mouth 3-5 days a week.
* Participants will get pembrolizumab in a vein for 30 minutes 1 day each cycle.

Participants will keep a study medication diary.

During cycle 1, participants will have blood taken multiple times on days 1 and 2.

Every 3 cycles, participants will repeat screening tests.

Participants will have a mandatory tumor biopsy.

When they finish treatment, participants will have a physical exam and blood tests.

DETAILED DESCRIPTION:
Background:

* Non-small cell lung cancers (NSCLC) esophageal cancer (EsC) and malignant pleural mesotheliomas (MPM) account for approximately 185,000 deaths annually in the United States, with over two thirds of patients presenting with advanced, incurable disease. 1st-line platinum-based chemotherapy for advanced NSCLC, esophageal cancer (ESCs) or malignant pleural mesothelioma (MPM) produces transient responses at best, with most patients succumbing to disease within 12-16 months following diagnosis.
* Recent randomized clinical trials have demonstrated response rates approximating 20% in unselected patients with advanced NSCLC or EsC, and nearly 45% in patients with tumors exhibiting high level expression of programmed death ligand 1 (PD-L1) following administration of pembrolizumab, a humanized monoclonal anti-Programmed cell death protein 1 (PD-1) antibody.
* Approximately 17% of unselected MPM patients have exhibited objective responses following administration of pembrolizumab or other PD-1 inhibitors.
* Preclinical studies have demonstrated that epigenetic drugs such as deoxyribonucleic acid (DNA) demethylating agents and histone deacetylase (HDAC) inhibitors can prime cancer cells and tumor microenvironments thereby enhancing efficacy of immune checkpoint inhibitors.
* Although a potent DNA demethylating agent, Decitabine has poor bioavailability and inconsistent distribution in solid tumors due to rapid inactivation by cytidine deaminase (CDA) which is present in high levels in many organs.
* Recent studies in rodents and nonhuman primates, as well as a Phase 1 clinical trial (NCT#01685515) in patients with sickle cell disease have demonstrated that oral tetrahydrouridine (THU), an inhibitor of CDA, significantly enhances bioavailability/solid-tissue-distribution of low dose oral Decitabine (DAC), thereby enhancing systemic DNA demethylation with acceptable toxicities.
* Preliminary results of recent clinical trial suggest that oral DAC-THU can increase the frequency and magnitude of responses to immune checkpoint inhibitors in lung cancer patients with low or absent intra-tumoral PD-L1 expression.
* These data support further evaluation of oral DAC-THU in combination with immune checkpoint inhibitors for therapy of thoracic malignancies.

Objectives:

Phase I

-To define pharmacokinetics, toxicities and maximum tolerated dose of oral DAC-THU in combination with pembrolizumab in patients with inoperable, or unresectable locally advanced or metastatic NSCLC, EsC, or MPM.

Phase II

-To determine clinical response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria to oral DAC-THU in combination with pembrolizumab in patients with inoperable, or unresectable, locally advanced or metastatic NSCLC, EsC, or MPM.

Eligibility:

Inclusion Criteria

* Male or female, 18 years or older with histologically or cytologically proven, inoperable, or unresectable locally advanced, or metastatic NSCLC, EsC, or MPM.
* Measurable disease.
* Patients with high PD-L1 expression ((Bullet) 50%) and low PD-L1 expression (0-49%) in cancer cells by immunohistochemistry are eligible.
* NSCLC patients with no prior systemic treatment, or those with prior first line treatment including an immune checkpoint inhibitor are eligible for study.
* MPM patients who have received, refused, or are ineligible for first line chemotherapy are eligible.
* Patients with EsC including Seiwert-Stein Type I and Type II gastro-esophageal junction (GEJ) carcinomas who have received or refused standard of care first line therapy and/or targeted therapy are eligible.
* Patients who received DNA demethylating agents or PD-1/PD-L1 inhibitors for another malignancy may be eligible for study if there were no dose-limiting immune related events, and there has been either no clinical evidence of disease or minimal residual disease that has been stable for at least three years.
* Willingness to undergo tumor biopsies if safely accessible per PI discretion before and after treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 2.
* No evidence of unstable or decompensated myocardial disease; adequate pulmonary reserve.
* Adequate renal, hepatic and hematopoietic function.

Exclusion Criteria

* Patients with any targetable mutation for which there is approved first, or second line therapy.
* Serious cardiovascular conditions.
* Active Hepatitis A, Hepatitis B or Hepatitis C.
* Human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Other active infection requiring systemic therapy.
* Pregnant or breastfeeding women.
* Patients who are receiving systemic corticosteroids.
* Patients receiving another investigational agent.
* Another malignancy.

Design:

* The Phase I component will be a standard 3+3 design combining high and low PD-L1 expressers with incremental dose escalation of oral DAC-THU to define maximum tolerated dose (MTD).
* Simon 2-stage design for Phase II studies will be used to determine clinical response at the MTD.
* Patients will receive oral DAC-THU- on T-W for two weeks out of every 3 for 9 weeks
* Pembrolizumab will be administered on Wednesday, Thursday or Friday at a fixed intravenous dose of 200 mg every 3 weeks.
* One cycle is three weeks; one course is 9 weeks. Treatment evaluation using RECIST 1.1 every 10 +/- 1 weeks.
* Those patients exhibiting disease progression or unacceptable toxicities will be removed from study. Patients exhibiting stable disease or disease regression will be offered an additional course of therapy followed by treatment evaluation. Treatment will continue in this manner until off-study criteria have been met.
* Once the MTD for DAC/THU has been identified, the MTD dose level will be expanded by 4 patients to confirm its safety. Then, including these 10 patients at the MTD, a total of 10 NSCLC patients with high (50% or greater) intratumoral PD-L1 expression and 10 NSCLC patients with low (0-49%) intratumoral PD-L1 expression will be accrued to the first stage of each of two separate Phase II cohorts using individual Simon optimal designs. If 5 or more patients of the 10 first stage NSCLC patients in the high PD-L1 cohort respond to treatment, the cohort will be expanded to 23 patients. If 11 of 23 of these patients respond to treatment, the trial will be deemed positive for NSCLC with high PD-L1 expression. If 2 or more of the 10 first stage NSCLC patients in the low PD-L1 expression cohort respond to treatment, the cohort will be expanded to 29 patients. If 6 or more of these 29 patients experience a response, the trial will be deemed positive for NSCLC with low PD-L1 expression. Up to 10 EsC patients, including those considered to be part of the Phase I component after the MTD has been identified, will be enrolled into a separate cohort to examine responses to DAC-THU/pembrolizumab at the MTD. If 2 or more of these 10 EsC patients respond to treatment, these findings may warrant an amendment or a separate Phase II trial to determine response rates to DAC-THU/pembrolizumab in EsC patients. Similarly, if 2 or more of 10 MPM patients respond to treatment, these findings may warrant an amendment or a separate Phase II trial to determine response rates to DACTHU/pembrolizumab in MPM.
* Biopsies of index lesions will be obtained at baseline and at treatment evaluation following the first course of therapy for analysis of pharmacodynamic endpoints.
* Patients will be followed for toxicity for at least 30 days after treatment has been discontinued, start of new anti-cancer treatment or until death, whichever occurs first.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed, inoperable or unresectable, locally advanced, or metastatic non-small cell lung cancers (NSCLC) or esophageal cancers including Seiwert-Stein Type I and Type II gastro-esophageal junction (GEJ) carcinomas, or malignant pleural mesothelioma (MPM).
* NSCLC patients with no prior systemic treatment or those with prior first line treatment including an immune checkpoint inhibitor, are eligible for study.
* Patients with esophageal and gastro-esophageal junction (GEJ) cancers are potentially eligible for study if they have received or refused first line standard of care cytotoxic therapy, and subsequent targeted therapy if appropriate.
* Patients with MPM are eligible for study if they have received, refused or are ineligible for first line chemotherapy.
* Patients who received deoxyribonucleic acid (DNA) demethylating agents or Programmed cell death protein 1 (PD-1)/Programmed Cell Death Ligand 1 (PD-L1)/PD-L1 inhibitors for another malignancy may be eligible for study if there were no dose-limiting immune related events, and there has been either no clinical evidence of disease or minimal residual disease that has been stable for at least three years.
* Patients must have analysis of PD-L1 expression in cancer cells quantitated by immunohistochemistry analysis.

  * Patients in Cohort 1 (Dose Escalation) may have any level of expression.
  * Patients in Cohort 2 (Dose Expansion: NSCLC with high PD-L1) must have greater than or equal to 50% expression in cancer cells.
  * Patients in Cohort 3 (Dose Expansion: NSCLC with low PD-L1) must have 0-49% expression. Note: Patients in this cohort must have been offered and refused standard of care platinum-based chemotherapy
  * Patients in Cohort 4 (Dose Expansion: Esophageal carcinomas (ESCs)) may have any level of expression.
  * Patients in Cohort 5 (Dose Expansion: MPM) may have any level of expression.
* Measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Willingness to undergo tumor biopsies if safely accessible per principal investigator (PI) discretion before and after treatment.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of Decitabine (DAC) and Tetrahydrouridine (THU) in combination with Pembrolizumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* Patients must be without evidence of unstable or decompensated myocardial disease; and must have adequate pulmonary reserve evidenced by Forced expiratory volume in the first second (FEV1) and diffusing capacity of lung for carbon monoxide (DLCO) greater than or equal to 35% predicted; oxygen saturation equal to or greater than 90% on room air by pulse oximetry or arterial blood gas (ABG) (to be drawn if pulse oximetry < 90% on room air)
* No immunosuppressive medications except non-systemic corticosteroids
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL (without transfusion or cytokine support)
  * absolute lymphocyte count greater than or equal to 800/mcL
  * platelets greater than or equal to 100,000/mcL
  * Prothrombin time (PT) no more than 2 seconds above the upper limit of normal (ULN)
  * total bilirubin < 1.5 X institutional upper limit of normal OR direct bilirubin less than or equal to ULN for patients with total bilirubin > 1.5 ULN
  * serum albumin greater than or equal to 2.0 mg/dL
  * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase, (SGOT)/Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) less than or equal to 2.5 X institutional ULN
  * creatinine less than or equal to 1.6 mg/ml OR creatinine clearance (eGFR) greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal at the time DAC-THU and pembrolizumab treatment commences.
* Patients with history of brain metastases except those with meningeal carcinomatosis or leptomeningeal disease may be eligible for treatment a minimum of 1 week following completion of gamma knife or whole brain radiotherapy, or 4 weeks following surgical resection of brain metastasis provided post-treatment magnetic resonance (MR) scan reveals no evidence of active disease, and no ongoing need for systemic steroids.
* Patients with laboratory evidence of autoimmune disease (e.g., positive anti-nuclear antibodies (ANA) or lupus anticoagulant) without associated symptoms; vitiligo, or mild autoimmunity not impacting the function of organs, such as Hashimoto or psoriasis may be eligible for study.
* The effects of DAC-THU and pembrolizumab on the developing human fetus are unknown. For this reason and because antineoplastic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men who engage in sexual activity must agree to use 2 forms of contraception at least 1 of which must be highly effective (intrauterine device [IUD], hormonal, tubal ligation; not highly effective includes barrier method) prior to study entry, for the duration of study participation and for 60 days after completion of the study treatment. Should a woman become pregnant, or suspect she is pregnant, while she or her partner is participating in this study the study participant should inform the study physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients with cancers harboring any targetable mutation for which there is approved first, or second line therapy, unless standard care of therapy refused.
* Clinically significant cardiovascular / cerebrovascular disease as follows: cerebral vascular accident / stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class greater than or equal to II), serious cardiac arrhythmia, clinically significant bleeding or clinically significant pulmonary embolism
* Active Hepatitis A, Hepatitis B (e.g., HB surface antigen (sAg) reactive) or Hepatitis C virus (e.g., HCV ribonucleic acid (RNA [qualitative] is detected).
* Human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness due to unknown effects of DAC-THU on systemic immunity.
* Other active infection requiring systemic therapy.
* Pregnant women are excluded from this study because DAC-THU may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DACTHU, breastfeeding should be discontinued if the mother is treated with DAC-THU. These potential risks may also apply to other agents used in this study.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Patients who are receiving systemic corticosteroids.
* Patients with history of or active autoimmune disease including thyroiditis, colitis, nephritis, neuropathy or pneumonitis.
* Patients receiving another investigational agent.
* An additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in-situ cervical or anal cancer, or ductal carcinoma in-situ.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Thrombocytosis defined as platelet count >1,200,000/mcL.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the Database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0140.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT): Phase 1, Arm 1, Dose Escalation, ORIGINAL Dose Level 1: Participants received Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) q week with Pembrolizumab infusion q3weeks
- Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT): Phase 1, Arm 1, Dose Escalation, ORIGINAL Dose Level -1: Participants received Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) q week. Participants received Pembrolizumab infusion q3weeks.
- Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks: Phase 1, Arm 1, Dose Escalation, Revised Dose Level 1. Participants received Decitabine 0.21 mg/kg + Tetrahydrouridine 10mg/kg TW weekly x 2 weeks q 3 weeks. Participants received pembrolizumab infusion q 3weeks.
- Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks: Phase 1, Arm 1, Dose Escalation, Revised Dose Level -1. Participants received Decitabine 0.17 mg/kg + Tetrahydrouridine 10mg/kg TW weekly x 2 weeks q 3 weeks. Participants received pembrolizumab infusion q 3weeks.
- Enrolled to Revised Dose Level 1 But Not Treated: Participants who were enrolled but not treated.
Period: Phase I Dose Escalation
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Enrolled to Revised Dose Level 1 But Not Treated
Started | 2 | 2 | 4 | 0 (No participants were enrolled in this Arm/Group.) | 1
Completed | 1 | 1 | 1 | 0 | 0
Not Completed | 1 | 1 | 3 | 0 | 1
Not completed — Removed from protocol prior to treatment due to rapidly progressive esophageal obstruction. | 0 | 0 | 0 | 0 | 1
Not completed — Best interest of participant | 1 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Delay >3 weeks on treatment | 0 | 0 | 1 | 0 | 0
Period: Phase II Dose Expansion
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Enrolled to Revised Dose Level 1 But Not Treated
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled on Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Enrolled to Revised Dose Level 1 But Not Treated | Total
Number analyzed (Participants) | 2 | 2 | 4 | 0 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  | 0 | 0
  Between 18 and 65 years | 1 | 0 | 4 |  | 1 | 6
  >=65 years | 1 | 2 | 0 |  | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.74) | 80.85 (11.53) | 49.62 (10.02) |  | 62.4 (0) | 59.9 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 |  | 0 | 4
  Male | 0 | 1 | 3 |  | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 |  | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 3 |  | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 |  | 0 | 1
  Asian | 0 | 1 | 0 |  | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0 | 0
  Black or African American | 1 | 0 | 1 |  | 0 | 2
  White | 1 | 1 | 2 |  | 1 | 5
  More than one race | 0 | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4 |  | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate was measured using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 to determine if the combination of decitabine and tetrahydrouridine is associated with a response rate which exceeds that of Pembrolizumab alone in participants who have programmed death-ligand 1 (PD-L1) expression of at least 50% and those who do not. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Every 10 weeks (± 1 week) until disease progression or unacceptable toxicity or off study criteria is met. Longest participant on study 11 months.
Population: 1/9 participants did not receive any therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 2 | 2 | 4
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 0 | 0 | 1
  Progressive Disease | 0 | 1 | 1
  Unevaluable for response | 2 | 1 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Decitabine
Description: Maximum Tolerated Dose (MTD) is the maximum dose at which fewer than one-third of participants experience dose limiting toxicity (DLT) within the first 6 weeks (two cycles) of decitabine and tetrahydrouridine therapy. If one of three patients at any given dose level experiences DLT, up to three additional patients will be treated at this dose level. If only one of six patients exhibit DLT, subsequent patients will be enrolled into the next higher dose level. As soon as two patients at any given dose level develop DLT, no additional patients will be entered at that level. Subsequent patients will be accrued into the preceding dose level; if DLT is observed in less than two of six patients treated at this lower level, this dose will represent maximum tolerated dose (MTD). A DLT is any Grade 3 or greater toxicity that cannot be attributed to a cause other than study treatment during the first two cycles of Course 1 of therapy such as disease progression or intercurrent illness.
Time Frame: Within the first 6 weeks (two cycles)
Population: 1/9 participants did not receive any therapy.
Measure: Number; unit: mg/kg
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 2 | 2 | 4
mg/kg | NA — MTD was not found due to the termination of the study. | NA — MTD was not found due to the termination of the study. | NA — MTD was not found due to the termination of the study.

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Tetrahydrouridine
Description: as for outcome 2
Time Frame: Within the first 6 weeks (two cycles)
Population: Within the first 6 weeks (two cycles)
Measure: Number; unit: mg/kg
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 2 | 2 | 4
mg/kg | NA — MTD was not found due to the termination of the study. | NA — MTD was not found due to the termination of the study. | NA — MTD was not found due to the termination of the study.

4. Secondary Outcome: Changes in Circulating Tumor Cells (CTCs)
Description: Peripheral blood will be collected to correlate changes in circulating tumor cells with clinical response. CTCs will be assessed using ferrofluidic enrichment and multi-parameter flow cytometric detection. Baseline and post-treatment specimen collection after one course of therapy (Week 10 +/- one week).
Time Frame: Baseline and post-treatment after one course of therapy (Week 10 +/- one week)
Population: This outcome measure was not evaluated and was to be performed in bulk. No assays were performed due to the pandemic. Participants could not travel to the National Institutes of Health (NIH) to have samples drawn.
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Changes in Immune Cell Subsets in Peripheral Blood Mononuclear Cells (PBMC)
Description: Peripheral blood mononuclear cells (PBMC) will be assessed using multiparameter flow cytometry for immune subsets including but not necessarily limited to Tregs, myeloid-derived suppressor cells (MDSC), effector and exhausted cluster of differentiation 4 (CD4+), cytotoxic T lymphocytes (CD8+) T cells, and cluster of differentiation 14 (CD14 +) monocytes. Assessment will include functional markers, i.e., programmed cell death protein 1 (PD-1), programmed death-ligand 1 (PD-L1), T-cell immunoglobulin mucin-3 (TIM-3), cluster of differentiation 152 (CTLA-4), human leukocyte antigen (HLA) membrane heterodimeric glycoproteins (-DR) and/or cluster of differentiation 40 (CD40). Baseline and post-treatment specimen collection after one course of therapy (Week 10 +/- one week).
Time Frame: Baseline and post-treatment after one course of therapy (Week 10 +/- one week)
Population: as for outcome 4
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percent Viable Tumor Cells
Description: Portions of biopsy materials will be sent for frozen section or permanent section confirmation of malignancy, i.e., non-small cell lung cancers (NSCLC), esophageal carcinomas (Esc), malignant pleural mesothelioma (MPM) cells, and percent viable tumor cells. All of the analyses are predicated on acquisition of sufficient materials.
Time Frame: Baseline and post-treatment after one course of therapy (Week 10 +/- one week)
Population: This outcome measure was not done because 1 participant declined biopsy due to the pandemic. And one participant did not have adequate tissue to evaluate. All other participants did not have biopsies.
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Changes in Gene, Endogenous Retroviral (ERV), Micro Ribonucleic Acid (RNA) Expressions, Deoxyribonucleic Acid (DNA) Methylation Signatures and Tumor Microenvironment
Description: Tissue will be processed for focused gene, endogenous retroviral and microRNA expressions, and DNA methylation signatures using quantitative reverse-transcription polymerase chain reaction (RT-PCR), nanostring, pyrosequencing and digital droplet PCR techniques. Isolate serum for focused methylation analysis. If sufficient tissue is available, another portion will be imbedded in paraffin for subsequent immunostaining experiments, focusing on expression of genes focusing on those proteins encoded by genes that have been identified to be clearly activated by epigenetic therapy. If sufficient materials are present, additional more comprehensive analyses including multiplex immunohistochemistry analysis of tumor microenvironment may be performed with the focus of materials from participants treated at the maximum tolerated dose. All of the analyses are predicated on acquisition of sufficient materials.
Time Frame: Baseline and post-treatment after one course of therapy (Week 10 +/- one week)
Population: as for outcome 6
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 2 months/10 days, 10 months/29 days, 20 months/30 days for the first, second and third group respectively.
Population: 1/9 participants did not receive any therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 2 | 2 | 4
Participants | 2 | 2 | 4

9. Other Pre Specified Outcome: Number of Participants With a Dose Limiting Hematologic Toxicity (DLT)
Description: A DLT is any Grade 3 (severe) or greater toxicity that cannot be attributed to a cause other than study treatment during the first two cycles of Course 1 of therapy such as disease progression or intercurrent illness.
Time Frame: First two cycles of Course 1 of therapy
Population: 1/9 participants did not receive any therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
Number analyzed (Participants) | 2 | 2 | 4
Participants | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 2 months/10 days, 10 months/29 days, 20 months/30 days for the first, second and third group respectively.
Description: 1/9 participants did not receive any therapy.
Arm/Group | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks | Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 2/4 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) (N=2) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) (N=2) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks (N=4) | Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (1) | 1 (5) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Sunday, Monday, Tuesday (SuMT) (N=2) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Monday-Tuesday (MT) (N=2) | Decitabine 0.2mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks (N=4) | Decitabine 0.17mg/kg + Tetrahydrouridine 10mg/kg Every (q) Tuesday,Wednesday (TW) x 2 Weeks q3Weeks (N=0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (16) | 2 (23) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (9) | 2 (4) | 1 (11) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (6) | 2 (5) | 1 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03233724/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03233724/ICF_001.pdf